CLINICAL TRIAL: NCT03089060
Title: Clinical Trial on the Semi-occlusive Treatment of Traumatic Substance Defects of the Fingertip in Children and Adults With a Novel Silicone Finger Cap. ("Klinische Prüfung Zur Semiokklusiven Behandlung Von Traumatischen Substanzdefekten im Bereich Der Fingerendglieder Mittels Silikonfingerorthesen (Silikonfingelingen) Bei Kindern Und Erwachsenen")
Brief Title: Silicone Finger Cap ("Silikonfingerling")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopädie- und Rehatechnik Dresden GmbH (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORD0001/2014
Record Dates: First submitted 2017-03-07; First posted 2017-03-24 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Finger Injuries
Keywords: Fingertip Amputation; Fingertip Regeneration; Infection; Occlusive Dressings; Pediatric Surgery; Silicone Finger Cap
MeSH Terms: conditions — Finger Injuries; Infections

STUDY DESIGN:
Intervention Model Description: monocentric, prospective, randomized, controlled, pseudo-cross-over
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone Finger Cap (Experimental): Patients randomized to this arm will be treated with the novel silicone finger cap for the first two weeks of treatment.
  Interventions: Device: Silicone Finger cap; Device: Film Dressing
- Film dressing (Active Comparator): Patients randomized to this arm will be treated with conventional film dressings for the first two weeks of treatment.
  Interventions: Device: Silicone Finger cap; Device: Film Dressing

INTERVENTIONS:
Device: Silicone Finger cap — Treatment with silicone finger cap
Device: Film Dressing — Treatment with conventional film dressing

SUMMARY:
Amputation injuries of the fingertip are common in all ages. For decades it is known that conservatively treated fingertips can regenerate skin and soft tissues to form a functionally and cosmetically excellent new fingertip. Unfortunately, little is known about the mechanisms controlling this ability that, in humans, is confined to the fingertips. Even less is known about the bacteria that regularly colonize these wounds without noticeable negative impact on regeneration and healing. Medical evidence on fingertip regeneration in humans is largely limited to retrospective studies and case reports. This study will be the first randomized controlled trial on the conservative treatment of fingertip amputations in children and adults.

When managed without surgery, self-adhesive polyurethane film dressings are commonly used to establish a wet chamber around the injury. This provides the best conditions for tissue regeneration inhibiting the formation of scar tissue at the same time. Unfortunately these dressings do not offer mechanical protection, they do not stick to wet skin and leak malodorous wound fluid. The investigators therefore developed a silicone finger cap that deals with these problems offering a mechanically protected, wet chamber around the injury for optimal regeneration conditions. This finger cap also offers a puncturable reservoir for excess wound fluid, which by this route can be routinely analyzed for diagnostic and research purposes.

This randomized controlled trial will for the first time test acceptance, safety and efficacy of this novel medical device in comparison with conventional self-adhesive film dressings while gathering information on the clinical course and outcome of conservatively treated fingertip amputation injuries.

Based on sample size calculations for primary outcome, 22 patients older than 2 years will be enrolled within 24 hours after having suffered an injury distal to the distal interphalangeal joint comprising all layers of the skin with a substance defect that cannot be primarily adapted without further shortening of the finger or plastic surgery. Participants are randomly assigned to start their treatment for the first two weeks either with a conventional film dressing or with the novel silicone finger cap. They will be changed to the other modality for another two weeks before the patient or the guardian can decide, if they would want the film dressing or the finger cap for the rest of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* full skin substances defects distal to the distal interphalangeal joint (DIP-joint) unsuitable for primary surgical closure without further substance loss
* no more than five fingers per patient may be injured
* circumference of the proximal phalanx in between 3.0 cm and 9.0 cm
* signed informed consent

Exclusion Criteria:

* known hypersensitivity against medical silicone or self-adhesive films
* bony injuries requiring a surgical intervention
* bite injuries
* chronic dermatologic disorders of the hand
* intake of medications affecting wound healing, for instance/such as systemic (non-inhalative) glucocorticoids, immunosuppressive or blood-thinning medications
* known wound healing disorders
* ongoing or recently finished chemotherapy
* primary/congenital immunodeficiency
* diabetes mellitus
* pregnant or breastfeeding patients/women, as well as any women, when a pregnancy at the beginning or during the course of the study cannot be excluded (i.e. post-menopausal, oophorectomy or hysterectomy, contraceptive method with pearl index less than 1 %, sexual abstinence or partner with vasectomy)
* addiction or other diseases, which do not allow to assess the entity, scope and possible consequences of this clinical trial
* not cooperative patients
* participation in a clinical trial within the last four weeks

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Acceptance | At day 28 after injury
  Acceptance of the silicone finger cap in comparison with conventional film dressings. Patient decides which dressing he or she prefers for the remaining treatment.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | At Day 0, 1, 7, 14, 21, 28, 35, 42 resp. till wound healing is complete.
  Safety of the finger cap in comparison to the film dressing. Patients are asked for adverse events (AE) or serious adverse events (SAE).
Disease-specific quality of life | At Day 0, 1, 7, 14, 21, 28, 35, 42 and 4 months resp. till wound healing is complete.
  Determination of disease-specific quality of life during the treatment with the silicon finger cap in comparison to the film dressing using a modified quality of life Wuerzburg Wound Score
Unplanned dressing changes as measured by number of dressing changes in addition to number of visits according to study protocol. | Up to 42 days resp. till wound healing is complete.
  Necessity of unplanned dressing changes in comparison to the film dressing.
Microbiological colonization | At Day 0, 1, 7, 14, 21, 28, 35, 42 resp. till wound healing is complete (if wound fluid is aspirable).
  Changes in microbiological colonization in the wound during treatment using microbiological analysis.
Re-epithelialization rate | At Day 14, 28, 42 resp. till wound healing is complete.
  Measuring of re-epithelialization rate
Tissue growth | At day 28 and 4 months.
  Determination of tissue growth during treatment using medical ultrasound
Function of the regenerated perspiratory glands | At 4 months (Day 122).
  Ceck of function of the regenerated perspiratory glands using Moberg's Ninhydrin test.
Sensibility/Sensitivity of the injured fingertip | At 4 months (Day 122).
  Check of sensibility/sensitivity of the injured fingertip using 2-point-discrimination threshold in the area of the injury is checked in comparison to the corresponding finger of the contralateral hand
Cosmetic aspects, measured using a check list/questionnaire | At 4 months (Day 122).
  Checking a list of common deformities i.e. scarring, split nails.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fitze, Prof. Dr., Study Director — Technical University Dresden
Locations (1):
- University Hospital Carl Gustav Carus, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schultz J, Patel PA, Aires R, Wissing L, Glatte P, Seifert M, Gentzel M, Fitze G, Doyle AM, Sandoval-Guzman T. Human fingertip regeneration follows clinical phases with distinct proteomic signatures. NPJ Regen Med. 2025 Nov 5;10(1):51. doi: 10.1038/s41536-025-00441-y. PMID 41193504
- [Derived] Schultz J, Leupold S, Grahlert X, Pfeiffer R, Schwanebeck U, Schrottner P, Djawid B, Artsimovich W, Kozak K, Fitze G. Study protocol for a randomized controlled pilot-trial on the semiocclusive treatment of fingertip amputation injuries using a novel finger cap. Medicine (Baltimore). 2017 Oct;96(41):e8224. doi: 10.1097/MD.0000000000008224. PMID 29019891